CLINICAL TRIAL: NCT06164184
Title: Interest of the Cone Beam Scanner of Temporal Bones in the Analysis of Conductive Hearing Loss
Acronym: Cone-Beam
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8012
Record Dates: First submitted 2022-11-29; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Conductive Hearing Loss
Keywords: Conductive Hearing Loss; Cone Beam; Cone beam CT; CBCT; Temporal bones
MeSH Terms: conditions — Hearing Loss, Conductive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Conductive hearing loss is very common and the incidence increases with age. Until now, the scanner was the reference examination in the etiological diagnosis of deafness.

When performing a CT scan of temporal bones for the etiological diagnosis of conductive hearing loss, the quality of the image depends on the scanner brand and the acquisition parameters.

The investigators wish to show the usefulness of the cone beam in the diagnosis of conductive hearing loss

ELIGIBILITY:
Inclusion Criteria:

* Major subject (≥18 years old)
* Subject having performed a CT scan or a cone beam for pre- and post-operative conductive hearing loss between January 01, 2018 and December 31, 2020
* Subject who has not expressed his opposition, after being informed, to the reuse of his data for the purposes of this research.

Exclusion Criteria:

* Subject who expressed their opposition to participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major subject (≥18 years old) having performed a CT scan or a cone beam for pre- and post-operative conductive hearing loss between January 01, 2018 and December 31, 2020
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Show retrospectively that the superiority of the cone beam over the scanner in the diagnosis of conductive hearing loss | Files analysed retrospectively from January 01, 2018 to December 31, 2020 will be examined
  This superiority is based on the quality of the images allowing the visualization of the different elements of the middle and inner ears:
  Ossicles, windows, nerves (VII and VIII), cochlea, labyrinth

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Radiologie 1 - CHU de Strasbourg - France, Strasbourg, France